CLINICAL TRIAL: NCT06279936
Title: Neurobiological Underpinnings of Neuropsychological Consequences in Long COVID: Exploration of Two Translational Pathways
Brief Title: Neurobiological Underpinnings of Neuropsychological Consequences in Long COVID
Acronym: Cov-N-Psy
Status: Active, not recruiting | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: UZA Foundation (Unknown)
Responsible Party: Principal Investigator, Dr Livia De Picker, Clinical Professor, Universiteit Antwerpen
Other Study IDs: B3002021000171
Record Dates: First submitted 2024-02-08; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Long COVID
Keywords: brain fog; neuropsychological; depression; anxiety; immunological markers; cortisol
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Long Covid patients: Long Covid patients with (neuro)psychological complaints
  Interventions: Other: Neuropsychological battery; Other: Surveys and symptom severity questionnaires; Other: Blood withdrawal; Other: Saliva swabs
- Covid controls (Ca): COVID-19 survivors without persistent complaints
  Interventions: Other: Neuropsychological battery; Other: Surveys and symptom severity questionnaires; Other: Blood withdrawal; Other: Saliva swabs
- Non-Covid controls (Cb): healthy uninfected controls
  Interventions: Other: Surveys and symptom severity questionnaires; Other: Blood withdrawal; Other: Saliva swabs

INTERVENTIONS:
Other: Neuropsychological battery — COVID-19 patients with persistent complaints of cognitive disabilities (more than 4 weeks post-infection) in daily life are examined with an extensive neuropsychological test battery (see below) at the outpatient clinic of the University Psychiatric Centre in Duffel and at the University Hospital Antwerp. This battery covers a broad range of reliable and valid tests divided into six cognitive domains: attention, memory, visuospatial functions, language, executive functions and psychomotor speed/coordination. The neuropsychological examination lasts an average of 2 hours per participant. The tests are carried out by the same experienced neuropsychologist and also follow a standardized sequence. In addition to the neuropsychological assessment, two self-report scales are filled out by each patient. These scales are used to detect possible complaints of fatigue and possible cognitive problems which are experienced by the patient during daily life activities.
  Groups: Covid controls (Ca); Long Covid patients
Other: Surveys and symptom severity questionnaires — Both self-rated surveys and clinician administered questionnaires
Other: Blood withdrawal — Blood samples will be collected in a standardized manner by venipuncture. Two blood vials will be collected and processed to perform the following analyses:
  * serum collection tube(s) allowing for HERV-W ENV and serological assays
  * plasma collection tubes for the assessment of other immune-related biomarkers (including but not limited to CRP, IL-6, IL-1b, TNF-a, IFN-g, tryptophan, kynurenine, 3-OH-kynurenine, quinolinic acid, kynurenic acid, enzymes of the kynurenine pathway).
Other: Saliva swabs — Salivary cortisol measures will be used as functional measure of the HPA axis activity, as the unbound cortisol fraction in saliva is highly correlated to plasma cortisol. Baseline diurnal cortisol and CAR levels will be measured using saliva, collected at home with Salivette® (Sarstedt) synthetic swabs. The rationale behind the choice of home sampling, is to maximize normal circumstances and to minimize stress related to the measuring procedure.

SUMMARY:
Objectives:

To describe the standardized evaluation of the psychological and cognitive function of long COVID patients and their evolution, to compare immunological and HPA-axis related biomarkers between long COVID patients and healthy controls, to explore cross-sectional and longitudinal associations between immunological measures and long COVID symptoms.

Study design:

Cov-N-Psy is a longitudinal observational study. Three groups will be included from 2021 until 2023: long COVID patients with neuropsychological complaints (P), COVID-survivors without persistent complaints (Ca) and healthy volunteers without a history of COVID-19 (Cb). The total sample size is estimated on 130. Four visits are organized: at baseline, three, six and twelve months.

The study is organized in three work packages (WP). WP1 includes a blood withdrawal and psychometric questionnaires and is part of every visit. WP2 includes cortisol measurement in saliva and takes place on the baseline visit for every participant and on the third visit for patients. Finally, WP3 includes a neurocognitive assessment at baseline for patients and Ca controls and on the third visit for patients.

DETAILED DESCRIPTION:
Research Objectives

Describe the standardized evaluation of the psychopathological and neurocognitive function of long COVID NP patients and their evolution over time; Compare the immunological profile and the cortisol awakening response (CAR) of long COVID NP patients to those of COVID-19 survivors without persistent complaints and healthy uninfected controls; Explore the cross-sectional and longitudinal association between long COVID NP symptoms and immunological and cortisol measures.

Methodology

Recruitment and study population

Inclusion criteria - patients:

All patients 18-70 years referred to the University Psychiatric Hospital (Campus UZA and Campus Duffel) for psychological and/or cognitive complaints at least >4 weeks following a confirmed diagnosis of COVID-19 infection with a positive PCR test or an antibodies test will be invited to participate in the study. The sample size of the patients is estimated on 50 participants. The patients have to be examined by their treating physician before enrollment to make sure other medical causes for their complaints are excluded. A positive score on at least two domains (psychological /cognitive) is necessary during the screening phase.

Inclusion criteria - controls:

Two control groups, one of 30 healthy uninfected controls (Cb), another of 50 COVID-19 survivors without persistent complaints (Ca), matched on age, sex and education with the patient group will be included. The participants for Ca will be recruited in UZA and by advertising. The healthy controls (Cb) will be recruited by mailing within the hospital and by advertising. A positive score on maximum one domain (psychological / cognitive) is allowed in the absence of a psychiatric diagnosis (confirmed by the MINI) and when the complaint causes significant distress (which is investigated during the screening phase).

Exclusion criteria for each subgroup:

* HPA subgroup: Participant is pregnant or breastfeeding / Participant receives hormonal replacement therapy (contraception is allowed) /Participant is treated with cortisol <4 weeks ago
* Neurocognitive assessment: IQ < 90 (screened with Raven Standard Progressive Matrices (Short Form) (RSPM-SF) / Participant takes sedative medication: benzodiazepines (Larger than the equivalent of diazepam 10mg per day, Last administration <8 hours prior to the neurocognitive test), new sedative antipsychotics/antidepressants (<4 weeks), other medication from DRUID class III (<4 weeks), last administration <8 hours prior to the neurocognitive tests, or causing significant sedation / Severe substance abuse (alcohol + drugs) / Pre-existing neurological diseases causing cognitive problems.

Study design This is a longitudinal study, which will be organized into three work packages (WP1, WP2 and WP3). Enrollment will continue for an estimated period of 24 months, depending on the time course of the epidemic curve. Last-patient-in is expected no later than November 1st, 2023. Patients will be referred mainly by the University Hospital of Antwerp (UZA) and enrolled at first visit to the University Psychiatric Hospital (UPCD), where follow-up will also take place at 3, 6 and 12 months. Patients can also be referred by the Flemish long COVID patient support group.

WP1 includes a blood withdrawal and psychometric questionnaires and is part of every visit. WP2 includes cortisol measurement in saliva and takes place on the baseline visit for every participant and on the third visit for patients. Finally, WP3 includes a neurocognitive assessment at baseline for patients and Ca controls and on the third visit for patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria - patients:

* 18-70 years
* Diagnosis of long COVID
* (Neuro)psychological symptoms >4 weeks after infection
* Infection with SARS-Cov-2 was detected with PCR (or antigen test)
* Other causes for their complaints are excluded by their GP or specialist
* Positive score on at least 2 NP domains during the screening phase

Inclusion criteria - control a:

* 18-70 years
* No prolonged symptoms due to SARS-CoV-2 infection within 4 weeks after infection
* No current (Neuro)psychological symptoms
* Infection with SARS-Cov-2 was detected with PCR (or antigen test)
* A positive score on maximum one domain (psychological / cognitive) is allowed in the absence of a psychiatric diagnosis (confirmed by the MINI) and when the complaint causes significant distress (which is investigated during the screening phase).

Inclusion criteria - control b:

* 18-70 years
* No (known) infection with SARS-CoV-2
* No current or previous (neuro)psychological symptoms

Exclusion Criteria:

* General exclusion criteria:

Participant is unable to read and understand the consent form and patient-reported outcomes, complete study-related procedures, or communicate with the study staff and informed consent cannot realistically be obtained in retrospect or with the help of a competent family member or legal representative.

Exclusion criteria for each subgroup:

* HPA subgroup

  * Participant is pregnant or breastfeeding
  * Participant receives hormonal replacement therapy (contraception is allowed).
  * Participant is treated with cortisol <4 weeks ago
* Neurocognitive assessment:

  * IQ < 90 (screened with Raven Standard Progressive Matrices (Short Form) (RSPM-SF) (39)
  * Participant takes sedative medication
* Benzodiazepines: Larger than the equivalent of diazepam 10mg per day. Last administration <8 hours prior to the neurocognitive tests.
* New sedative antipsychotics/antidepressants (<4 weeks)
* Other medication from DRUID class III (<4 weeks), last administration <8 hours prior to the neurocognitive tests, or causing significant sedation.

  * Severe substance abuse (alcohol + drugs)
  * Pre-existing neurological diseases that influence cognitive functioning

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three participant groups will be included: 1) long COVID patients with neuropsychological complaints (P), 2) COVID-survivors without persistent complaints (Ca) and 3) healthy volunteers (Cb).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of immunological and HPA-axis markers | Baseline (11/2021-12/2023) - FU (01/2022-12/2024)
  Compare the immunological profile and the cortisol awakening response (CAR) of long COVID NP patients to those of COVID-19 survivors without persistent complaints and healthy uninfected controls

SECONDARY OUTCOMES:
Rate of psychopathological and neurocognitive function of long COVID patients with neuropsychiatric complaints | Baseline (11/2021-12/2023) - FU (01/2022-12/2024)
  Describe the standardized evaluation of the psychopathological and neurocognitive function of long COVID NP patients and their evolution over time;
Cross-sectional and longitudinal association between long COVID NP symptoms (BDI, HDRS, STAI, ISI, KEDS, FSS, NP battery ...) and immunological and cortisol measures (CAR, cytokines, serology, WBC, CRP, mitochondrial markers, TRYCATS, ...) | Baseline (11/2021-12/2023) - FU (01/2022-12/2024)

CONTACTS AND LOCATIONS:
Locations (1):
- SINAPS, Duffel, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.sinapsduffel.com/longcovid

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT06279936/Prot_SAP_000.pdf